CLINICAL TRIAL: NCT00481988
Title: Randomized, Double Blind Crossover Study of the Treatment of Major Depressive Episode With Transcranial Direct Current Stimulation (tDCS)
Brief Title: Treating Depression With Transcranial Direct Current Stimulation (tDCS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5405
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Depression
Keywords: depression; transcranial direct current stimulation; direct current stimulation; tdcs
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- transcranial direct current stimulation (Active Comparator): The active group of patients will receive active Iomed II Phoresor transcranial direct current stimulation for the first two weeks followed by another two weeks of active transcranial direct current stimulation.
  Interventions: Device: transcranial direct current stimulation
- sham tDCS (Sham Comparator): The patients in the sham arm receive active Iomed II Phoresor transcranial direct current stimulation for the second two weeks of the clinical trial only. For the first two weeks the Iomed II Phoresor constant current generator is turned on for 10 seconds to produce the tingling sensation on the scalp experienced by the patients in the active arm but the generator is then turned off and the patients receive no stimulation for the remainder of the 20 minute session.
  Interventions: Device: iomed phoresor transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Two damp sponges, one placed on the left side of the forehead, the other on the left arm. 0.1mA of current is passed for 20 minutes.
  Other Names: ioMed Phoresor
  Arms: transcranial direct current stimulation
Device: transcranial direct current stimulation — transcranial direct current stimulation delivers one milliamp of direct current, supplied by a constant current generator, the the left dorsolateral prefrontal cortex through a scalp electrode. The treatment is given for 20 minutes a day.
  Other Names: Phoresor II Auto model PM850
  Arms: transcranial direct current stimulation
Device: transcranial direct current stimulation — one milliamp of direct current applied to the left dorsolateral prefrontal cortex through a scalp electrode
  Other Names: Phoresor II Auto model PM850
  Arms: transcranial direct current stimulation
Device: iomed phoresor transcranial direct current stimulation — for the sham group the current is turned off after 10 seconds
  Other Names: phoresor II auto model PM850
  Arms: sham tDCS

SUMMARY:
The purpose of this study is to see if transcranial direct current stimulation may improve the symptoms of depression.

DETAILED DESCRIPTION:
The purpose of this study is to learn about a brain stimulating procedure called transcranial direct current stimulation (tDCS). In tDCS therapy, two moistened sponges are applied to the forehead while a small amount of electric current flows between them. These electrodes are placed on the head so that the electricity will pass through a region in the brain that is believed to contribute to depression. This study is intended to test the theory that the electromagnetic field created by the current may affect this region of the brain in a way that may improve the symptoms of depression. This may affect brain activity and function.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of a major depressive episode or bipolar disorder and is currently in a major depressive episode (without psychotic features)
* Total pretreatment HDRS (Hamilton Depression Rating Scale)-24 score >= 18 (The Hamilton Depression Rating Scale is an interviewer scored tool for assessing the severity of depressive symtoms. The scale ranges from 0 (no symptoms, absence of depression) to 64

Category Ham-24 Score Normal, not depressed 9 or less Mildly depressed 10 to 19 Moderately depressed 20 to 29 Markedly/severely depressed 30 or more)

* Capable and willing to provide informed consent

Exclusion Criteria:

* History of depression previously untreated with medication, bipolar disorder, schizophrenia, schizoaffective disorder (non mood disorder), psychosis, depression secondary to a medical condition, mental retardation, substance dependence or abuse within the past year (except nicotine), psychotic features in this or previous episodes, amnestic disorder, dementia or mms<24, DELIRIUM
* Significant current history of autoimmune, endocrine, viral or vascular disorder affecting the brain
* History of unstable cardiac disease, uncontrolled hypertension, or sleep apnea
* Changes in psychotropic medications within two weeks prior to study entry or patient is unable to maintain stable doses throughout the study trial
* Subject has an active suicidal plan and/or attempted suicide in the past twelve months
* Patients with a CGI of 6 or greater
* Subject is pregnant or has a positive pregnancy serum test

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Bulow, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] COSTAIN R, REDFEARN JW, LIPPOLD OC. A CONTROLLED TRIAL OF THE THERAPEUTIC EFFECT OF POLARIZATION OF THE BRAIN IN DEPRESSIVE ILLNESS. Br J Psychiatry. 1964 Nov;110:786-99. doi: 10.1192/bjp.110.469.786. No abstract available. PMID 14211695
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- See also: National Institute of Mental Health - Depression — http://www.nimh.nih.gov/publicat/depression.cfm
- See also: Study summary on the Brain Stimulation Division web site — http://www.brainstimulation.columbia.edu/research/clinical/depression.html#TDCS

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: 2006-2009 Location: community Approved sample size: 23 Total number of participants enrolled: 19
Pre-assignment Details: One patient was dropped by the investigator when he had a Hamilton Depression Rating Scale (HDRS) of 8 prior to baseline ratings (DRSS 20 is the minimum for inclusion in the study).
Groups:
- Iomed II Phoresor Transcranial Direct Current Stimulation: The active group of patients will receive active Iomed II Phoresor transcranial direct current stimulation for the first two weeks followed by another two weeks of active transcranial direct current stimulation.
- Sham Iomed II Phoresor Transcranial Direct Current Stimulation: The sham group receives sham stimulation for the first two weeks of the study followed by active treatment in the second two weeks. To mimic the sensation of active treatment and maintain the blind of the study, in the sham arm the Iomed II Phoresor constant current generator is turned on for 10 seconds to produce the tingling sensation on the scalp experienced by the patients in the active arm but the generator is then turned off and the patients receive no stimulation for the remainder of the 20 minute session.
Period: Overall Study
Arm/Group | Iomed II Phoresor Transcranial Direct Current Stimulation | Sham Iomed II Phoresor Transcranial Direct Current Stimulation
Started | 12 | 9 (one patient was dropped from the study before randomization)
Crossover | 11 (patient dropped out of study after 5 sessions to pursue other treatment options) | 8 (patient dropped out of study after 5 sessions to illness unrelated to study)
Completed | 11 | 8
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: One patient dropped out of study after 5 treatments due to One patient dropped out of study after 5 treatments to pursue other treatment options One patient dropped by investigator when patient had HDRS of 8 at baseline ratings One patient dropped out of study after 1 treatment to pursue other treatment options
Groups:
- Transcranial Direct Current Stimulation: one group of patients will receive active transcranial direct current stimulation for the first two weeks followed by another two weeks of active transcranial direct current stimulation, whereas the second group of patients will receive two weeks of sham transcranial direct current stimulation followed by two weeks of active transcranial direct current stimulation
- Sham tDCS: the constant current generator is turned on for 10 seconds to produce the tingling sensation on the scalp experienced by the patients in the active arm but the generator is then turned off and the patients receive no stimulation for the remainder of the 20 minute session.
- Total: Total of all reporting groups
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45 (2) | 45 (2) | 45 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (24 Question Version), a Standardized Assessment Tool for Measuring Severity of Depression Where 0 is the Minimum Score (no Depressive Symptoms) and 40 is the Maximum (Severe Depression).
Description: The Hamilton Rating Scale for Depression (HRS,24 question version), is a standardized assessment tool for measuring severity of depression where 0 is the minimum score (no depressive symptoms) and 40 is the maximum (severe depression).I am reporting the number of participants with stable remission which is defined as an HDRS < 10 for 2 weeks.
Time Frame: Two weeks
Population: 20 patients were enrolled in the study and 17 patients completed it. The 17 patients who completed the study are the population analyzed.
Measure: Number; unit: participants
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS
Number analyzed (Participants) | 9 | 8
participants | 2 | 2

2. Secondary Outcome: Beck Depression Inventory II
Description: patient self report of depressive symptoms
Time Frame: Two weeks
Population: Data for the secondary outcome measure was incompletely collected and not analyzed.
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/8
Other Adverse Events (participants affected / at risk) | 2/19 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Direct Current Stimulation (N=19) | Sham tDCS (N=8)
scalp burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — two of the participants suffered scalp burns under the site of the sponge electrode. These were similar to sunburns and resolved completely by the next day. These burns occurred only in subjects receiving active tDCS, not sham tDCS.

LIMITATIONS AND CAVEATS:
Data for the secondary outcome measure (Beck Depression Inventory) was incompletely collected and not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No